CLINICAL TRIAL: NCT01496404
Title: A Randomized Controlled Trial Comparing the Cosmetic Outcome of Electrocautery Versus Scalpel for Surgical Skin Incisions
Brief Title: Electrocautery Versus Scalpel for Skin Incisions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: St. Paul's Hospital, Canada (Other)
Responsible Party: Principal Investigator, Dr. Carl J Brown, Head, Division of General Surgery, Providence Health Care, St. Paul's Hospital, Canada
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: H11-02242
Record Dates: First submitted 2011-12-18; First posted 2011-12-21 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Wound Complication; Surgical Wound Infection; Post-operative Pain
Keywords: Electrocautery
MeSH Terms: conditions — Surgical Wound Infection; Pain, Postoperative | interventions — Electrocoagulation; Laser Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Electrocautery (Experimental): Epidermis and dermis incised with cutting setting of electrocautery.
  Interventions: Procedure: Electrocautery
- Scalpel (Active Comparator): Control, incision of epidermis and dermis with scalpel.
  Interventions: Procedure: Scalpel

INTERVENTIONS:
Procedure: Electrocautery — Electrocautery using cutting mode of epidermis and dermis of skin.
  Arms: Electrocautery
Procedure: Scalpel — Incising skin (epidermis and dermis) with scalpel.
  Arms: Scalpel

SUMMARY:
The aim of this research project is to compare electrocautery to scalpel for laparotomy skin incisions, with the following objectives:

1. To investigate whether electrocautery produces a cosmetically inferior surgical scar.
2. To compare the rates of wound infection with each technique.
3. To determine if electrocautery results in less postoperative pain. Our null hypothesis is that electrocautery is equivalent to scalpel for creating skin incisions; with respect to wound cosmesis, wound infection rate, and post-operative pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 19 years old
* bowel resection surgery
* incision is 3cm or larger

Exclusion Criteria:

* Diagnosed with a connective tissue disease (e.g. Systemic lupus, scleroderma, polymyositis, dermatomyositis, Marfan syndrome, Ehler's Danlos, etc.)
* The site of planned surgery has a previous surgical scar.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2012-01; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Scar Cosmesis | 6 months
  At 6 months post-operative, patients' scars will be evaluated by two independent trained blinded observers who will use the Patient Observer Scar Assessment Scale (POSAS) and the Vancouver Scar Scale (VSS) to evaluate the cosmesis of the surgical scar. Patients, who are blinded to the type of incision they have received, will also subjectively assign a score to their scar using the POSAS.

SECONDARY OUTCOMES:
Wound Infection Rate | within 6 months post-operatively
  Superficial incisional surgical site infection as defined by the Centres for Disease Control (CDC).
Post-operative wound pain | within 5 days post-operatively
  Patients will also be asked to record their daily post-operative incision pain using the visual analogue score (VAS) until post-operative day 5.

CONTACTS AND LOCATIONS:
Overall Officials: Carl J Brown, MD MSc FRCSC, Principal Investigator — Providence Health, University of British Columbia; Lisa NF Aird, BSc MD, Principal Investigator — University of British Columbia
Locations (1):
- St Paul's Hospital, Vancouver, British Columbia, Canada

REFERENCES:
- [Derived] Aird LN, Bristol SG, Phang PT, Raval MJ, Brown CJ. Randomized double-blind trial comparing the cosmetic outcome of cutting diathermy versus scalpel for skin incisions. Br J Surg. 2015 Apr;102(5):489-94. doi: 10.1002/bjs.9751. Epub 2015 Feb 18. PMID 25692789